CLINICAL TRIAL: NCT05980130
Title: RFCBT I - Proof of Concept Study/Single Subject Design
Brief Title: Can Rumination-Focused Cognitive Behavioral Therapy Reduce the Risk of Cardio-vascular Disease?
Acronym: RFCBT-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Patrick Possel, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23.0150
Record Dates: First submitted 2023-06-07; First posted 2023-08-07 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Rumination; Depressive Symptoms; Blood Pressure
Keywords: rumination; depressive symptoms; blood pressure; rumination-focused cognitive behavioral therapy; Proof of Concept Study; Single subject design
MeSH Terms: conditions — Rumination Syndrome; Depression

STUDY DESIGN:
Intervention Model Description: Single subject design
Masking Description: This is a Single subject design study. Thus, as all participants receive the intervention, there is no masking possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFCBT (Experimental): This is a single subject design study. Thus, all participants receive Rumination-Focused Cognitive Behavior Therapy
  Interventions: Behavioral: Rumination-Focused Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Rumination-Focused Cognitive Behavior Therapy — The RFCBT exclusively addresses one possible mechanism underlying depression, rumination. In general, a participant and their therapist will identify when the participant ruminates in an unhelpful manner, what triggers the rumination, what function the rumination fulfills for the participant, and how the participant already does to stop ruminating. Building on this knowledge both together will change the environment to reduce the likelihood of the participant to ruminate, use consciously strategies to stop rumination when it occurs, and replace rumination by more helpful strategies. In the proposed single subject study, the participant and the therapist will meet in person or using a UofL approved video platform up to 18 times for 50-minutes.

SUMMARY:
Many people know that a poor diet, exercise, smoking, and alcohol use cause heart disease. However, a less known factor that increases the risk of heart disease is depression. In addition, heart disease can also make depression worse. Almost half of American adults have some form of heart disease. Patients with low income are at an even greater risk. The circular relation between depression and heart disease raises the question of whether or not there are factors that lead to both. Attacking a factor that affects both depression and heart disease could help prevent them both. One such factor is rumination which is when someone tends to have repeated negative thoughts that loop without end. This loop in turn tears and wears down the body over time, making the person be at risk for heart disease and depression. Rumination-Focused Cognitive Behavioral Therapy (RFCBT) is a tool that targets rumination and, by doing so, reduces the risk for depression. While research has shown RFCBT helps to reduce or stop the loop that leads to depression, this project will further look at the effect of RFCBT on measures of heart health persons with low income.

DETAILED DESCRIPTION:
Objectives Objective #1: Determine whether RFCBT will impact blood pressure as a biomarker of cardiovascular health. The investigators hypothesize that RFCBT will lead to an improvement in blood pressure.

Objective #2: Determine whether RFCBT will impact stress biomarkers of cardiovascular health. The investigators hypothesize that RF-CBT will lead to an improvement of salivary cortisol.

Objective #3: Determine whether RFCBT will impact inflammatory biomarkers of cardiovascular health. The investigators hypothesize that RF-CBT will lead to an improvement of salivary C-Reactive Protein (h-CRP), interleukin (IL-6), and tumor necrosis factor-alpha (TNF-α).

Objective #4: Determine the acceptability of RFCBT for individuals with low income. While the investigators cannot predict the themes that will be generated, the information will have implications for the use of RFCBT with individuals with low income.

Study Design/Methodology The investigators will use a multiple baseline design - a type of Single Case Experimental Design (SCED) and collect survey, interview, and biological (blood pressure & saliva) data. Because of the study design, all participants will receive Rumination-Focused Cognitive Behavioral Training (RFCBT); the study is not blinded, and no non-intervention control group is necessary. As participants will be selected non-randomly, they will be randomly assigned to a group or in other words after how many weeks of baseline phase they will perceive RFCBT using the random number generator in the statistics package R. That is, 1/3rd of the participants will participate in 5 baseline waves of data collection, each one week apart, before starting RFCBT, another 1/3rd of participants will participate in 6 baseline waves before starting RFCBT, and the final 1/3rd of participants will participate in 6 baseline waves before starting RFCBT. Thus, all participants will participate in 5 to 7 weekly baseline waves. Next, each participant will participate with their trainer in up to 18 50-minute meetings of RFCBT. In this time, each participant will participate in 6 to 9 waves of training data collection (one wave of data collection every 2 RFCBT meetings). After completion of the training, each participant will be followed for another 10 weeks during which they participate in 5 waves of follow-up data collection (one wave of data collection every 2 weeks). Thus, each participant participates in 28 to 36 weeks in the study and takes part in 16 to 21 waves of data collection.

The investigators plan to recruit 27 adults with low income who have an elevated Response Style Questionnaire (RSQ)-Brooding score (>= 11), Patient Health Questionnaire (PHQ)-9 score (10-20), and blood pressure (systolic blood pressure [SBP]/ diastolic blood pressure [DBP]: >= 120 and/or 80) - that Have A Heart Clinic personnel administers regularly - and speak fluent English. There are no other exclusion criteria including any medical or psychological treatment. Patients who fulfill the above listed inclusion criteria are referred by Have A Heart Clinic personnel to the research team.

At each wave of data collection, the investigators will administer all the surveys listed in this report. All questions will be administered at each wave except for the questions about demographic information which will be asked during Baseline-1 only.

To measure blood pressure, the investigators will use an oscillometric measurement device. To do so, a blood pressure cuff will be placed about an inch above the elbow crease. For reliability purposes, blood pressure will be measured three-times with about 1 minute time between the measures.

To measure cortisol, h-CRP, IL-6, and TNF-α levels in saliva, participants will also be asked to provide saliva samples. Participants will be asked to avoid eating food or drinking caffeine for 3 hours prior to the saliva data collection in order to prepare for the saliva testing.

Once after the participants finish the RFCBT, they will be invited to take part in a semi-structured interview to explore their experiences in and acceptability of the training. The investigators intend to do these interviews with all participants who begin RFCBT (i.e., defined as completing at least one 50-minute meeting with their trainer), including those who drop out of the training, in-person, by phone, or a secure video platform.

The RFCBT exclusively addresses one possible mechanism underlying depression, rumination. In general, a participant and their trainer will identify when the participant ruminates in an unhelpful manner, what triggers the rumination, what function the rumination fulfills for the participant, and how the participant already does to stop ruminating. Building on this knowledge both together will change the environment to reduce the likelihood of the participant to ruminate, use consciously strategies to stop rumination when it occurs, and replace rumination by more helpful strategies. In the proposed single subject study, the participant and the trainer will meet in person or using a UofL approved video platform up to 18 times for 50-minutes.

Plan for Analysis of Results Following the best practice guidelines of the What Works Clearinghouse Standards for SCEDs, the investigators will examine consistency, intervention effect, immediacy, and auto-correlations for rumination, depressive symptoms, blood pressure, cortisol, h-CRP, IL-6, and TNF-α. The investigators will use Bayesian unknown changepoint models to estimate the parameters and model the treatment effect. A mixed effects model will be used to model the hierarchical structure of the data. The dependent variables are rumination, depressive symptoms, blood pressure, cortisol, h-CRP, IL-6, and TNF-α. The independent variable is phase. Bayesian estimation will be used to address the small sample nature of the data. For these statistical analyses the investigators will use R and "Just Another Gibbs Sampler" (JAGS). The investigators will conduct semi-structured interviews and analyze data using thematic analysis to generate themes associated with the data. The statistical program Dedoose will be utilized to facilitate this process.

ELIGIBILITY:
Inclusion Criteria:

* RSQ-Brooding score: >= 11
* PHQ-9 score: 10-20
* SBP: >= 120 and/or DBP: >= 80)
* fluent in English

Exclusion Criteria:

* None besides the described inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Response Style Questionnaire | Baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 1 week after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 2 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 3 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 4 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 5 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 6 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 7 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 9 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 11 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 13 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 15 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 17 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 19 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 21 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 23 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 25 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 27 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 29 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 31 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Response Style Questionnaire | 33 weeks after baseline 1
  sadness rumination, Score range: 5-20, higher score = more rumination
Patient Health Questionnaire-9 | Baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 1 week after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 2 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 3 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 4 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 5 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 6 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 7 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 9 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 11 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 13 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 15 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 17 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 19 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 21 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 23 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 25 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 27 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 29 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 31 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
Patient Health Questionnaire-9 | 33 weeks after baseline 1
  depressive symptoms, Score range: 0-27, higher score = more depressive symptoms
systolic blood pressure measures | Baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 1 week after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 2 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 3 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 4 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 5 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 6 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 7 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 9 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 11 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 13 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 15 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 17 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 19 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 21 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 23 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 25 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 27 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 29 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 31 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
systolic blood pressure measures | 33 weeks after baseline 1
  systolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | Baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 1 week after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 2 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 3 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 4 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 5 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 6 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 7 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 9 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 11 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 13 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 15 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 17 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 19 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 21 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 23 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 25 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 27 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 29 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 31 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure
diastolic blood pressure measures | 33 weeks after baseline 1
  diastolic blood pressure; score range: 0-200+, higher score = higher blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Possel, Dr.rer.soc., Principal Investigator — University of Louisville
Locations (1):
- Have a Heart clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No